CLINICAL TRIAL: NCT02073773
Title: Combinational Rehabilitative Therapy and Functional Brain Imaging for Patients Recovering From Motor Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore University of Technology and Design (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CIRB 2013/323/D
Record Dates: First submitted 2014-02-22; First posted 2014-02-27 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Ischaemic Stroke
Keywords: stroke, virtual reality based therapy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Levodopa; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual Reality based therapy, levodopa (Experimental): The VR therapy session consists of the subject interacting with a computer-based program in which they guide an avatar to gather items by using flexion and extension gestures of the affected upper limb. VR therapy sessions will last for 15-30 minutes depending on the subject's tolerance and participation. For patients who are unable to overcome gravity fully, they can still participate in this therapy by resting their arm on a table.
  Patients will receive a single dose of 100mg levodopa in combination with benserazide 2-3 hours before each additional Occupational therapy session or VR therapy session depending on the assigned group.
  Interventions: Drug: Levodopa; Other: Virtual Reality based therapy
- occupational therapy, levodopa (Active Comparator): The control group will receive and additional half an hour per working day of standard occupational therapy.
  Patients will receive a single dose of 100mg levodopa in combination with benserazide 2-3 hours before each additional Occupational therapy session or VR therapy session depending on the assigned group.
  Interventions: Drug: Levodopa

INTERVENTIONS:
Drug: Levodopa — Levodopa 100mg with benserazide 25mg will be administered 3 hours prior to the start of the daily PT/OT session to maximize its pharmacokinetic window ie. blood plasma levels in the narrow window during which functional rewiring of neural circuits is thought to occur.
  Levodopa at the lowest available dose (100mg P.O qd) has been shown to improve motor function of stroke patients and their corresponding quality of life. The treatment proposed can be incorporated into their daily rehabilitation routine. Early intervention (within 7-21 days of the infarct) raises the chance for neuroplasticity and improved recovery of their motor function in the short and long run. Levodopa has been proven to be safe to be used in stroke patients (Lancet. 2001 Sep 8;358(9284):787-90., Arch Phys Med Rehabil. 2008 Sep;89(9):1633-41.), however, the side effects of this medication may include nausea, unusual tiredness, dizziness, excessive watering of mouth.
  Other Names: Madopar
Other: Virtual Reality based therapy — The VR therapy session consists of the subject interacting with a computer-based program in which they guide an avatar to gather items by using flexion and extension gestures of the affected upper limb. VR therapy sessions will last for 15-30 minutes depending on the subject's tolerance and participation. For patients who are unable to overcome gravity fully, they can still participate in this therapy by resting their arm on a table.
  Arms: Virtual Reality based therapy, levodopa

SUMMARY:
The present proposal aims to assess whether a combined rehabilitation approach using virtual reality based therapy with motivational feedback, levodopa for pharmacotherapy and standard rehabilitative occupational therapy and physiotherapy will lead to signifcantly better outcomes for stroke recovery.

It is a randomised controlled trial with blinding of the assessors only. It will be preceeded by a Phase 1 pilot trial of the VR physiotherapy and standard therapy only. Recruited in-patient rehabilitation ward patients who have recently suffered stroke will be randomized, through a computer-based random number generator, to either one of two treatment arms:

1. Control occupational therapy + pharmacotherapy for 2 weeks
2. Assisted Virtual-Reality physiotherapy + pharmacotherapy for 2 weeks

DETAILED DESCRIPTION:
The study is designed as a single-blinded randomized controlled trial, preceeded by a Phase 1 pilot trial of the VR physiotherapy and standard therapy only.

Phase 1 will comprise of recruitment of up to 5 patients who have recently suffered a stroke who will be informed that they will receive ten 15- 30 minutes of VR therapy in addition to their standard stroke therapy. They will not receive any pharmacotherapy during this period. At the start and end of the VR phase, clinical assessment (Fugl-Meyer scores, Action Research Arm Test) will be made of each patient by a blinded clinician investigator.

From this data, calibration to the VR program will be made to ensure reproducibility of effectiveness of movements assessed.

Subsequently, for the main phase of the trial, recruited in-patients who have recently suffered stroke will be randomized, through a computer-based random number generator, to either one of two treatment arms:

1. Control occupational therapy + pharmacotherapy
2. Assisted Virtual-Reality physiotherapy + pharmacotherapy

Each patient will receive an initial functional Magnetic Resonace Imaging (fMRI) scan prior to the start of the study. The initial pilot single-centre study will be run in the Singapore General Hospital Rehabilitation Ward across a 2-week period, where participants will undergo daily 15-30 minute VR based therapy in addition to the physiotherapy/occupational therapy session they receive daily.

The VR therapy session consists of the subject interacting with a computer-based program in which they guide an avatar to gather items by using flexion and extension gestures of the affected upper limb. VR therapy sessions will last for 15-30 minutes depending on the subject's tolerance and participation. For patients who are unable to overcome gravity fully, they can still participate in this therapy by resting their arm on a table.

Patients will receive a single dose of 100mg levodopa in combination with benserazide 2-3 hours before an additional half an hour of occupational therapy to the weaker arm or VR therapy session, depending on the assigned group.

At the start and end of the trial, clinical assessment (Fugl-Meyer scores, Action Research Arm Test and Functional Independence Measure) will be made of each patient by a blinded clinician investigator. At the final (10th) session, patients will undergo the final fMRI scan. MRI scans will be analysed by blinded assessors.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-99yrs
* Right-handed
* Cognitively coherent, able to provide informed consent (MMSE >25)
* Newly diagnosed, first episode ischemic stroke in the past 2-21 days
* Motor score: Strength of 2-3 out of 5 on affected side upper limb

Exclusion Criteria:

* Declined consent to participate in the study
* Cognitive impairment or significant aphasia with inability to understand study requirements and inability to participate in therapy
* Other neurological or physical ailments with pre-existing motor weakness
* Haemorrhagic stroke
* Patient due to undergo significant medical interventions such as carotid endarthrectomy
* Patients on neuroactive agents prior to the stroke such as antidepressants
* Hypersensitivity to benserazide, levodopa, sympathomimetics, or any component of the formulation
* Use of MAO inhibitors within the last 14 days
* Patients with clinical or laboratory evidence of uncompensated cardiovascular, endocrine, renal, hepatic, hematologic, or pulmonary disease
* Patients with decompensated endocrine, renal, hepatic, cardiac disorders, psychiatric disorders, narrow-angle glaucoma, or closed-angle glaucoma;
* Patients <25 years of age (due to possibility of skeletal abnormalities from benserazide)
* Pregnancy or use in women of childbearing potential without adequate contraception.

Ages: 25 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Changes in the Fugl Meyer Upper Limb score at the start and end of the two weeks trial period | At the start and end of the 2 weeks period of trial therapy
  Fugl Meyer Upper Extremity Scale (FM) - a clinical assessment of upper limb tone, power and movement.

SECONDARY OUTCOMES:
Changes in the Action Research Arm Test (ARAT) | At the start and end of the 2 weeks period of trial therapy
  an assessment tool of upper limb grasp, grip, pinch and gross movement.
Changes in the Functional independence measure score | At the start and end of the 2 weeks therapy period
  An assessment of ability to perform 13 different activites of daily living and an assessment fo 5 measures of cognition necessary for independence

OTHER OUTCOMES:
Changes in Kinematic data of affected upper limb movement | At the start and end of the 2 weeks trial period
  The equipment used for the VR based therapy will record participant's joint angle displacement, hand path ratio and number fo repetitions completed
changes in resting state functional MRI imaging of the brain | At the start and end of the 2 weeks trial period
  fMRI imaging of the brain at the start and end of the trial period will assess changes in the area of brain activity that may be directly attributable to the effects of levodopa and rehabilitative therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Yee S NG, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, SIngapore, Singapore